CLINICAL TRIAL: NCT07290933
Title: Oral Food Processing for Digitally Constructed Complete Dentures Versus Conventional Complete Dentures: A Randomized Crossover Study
Brief Title: Oral Food Processing for Digitally Constructed Complete Dentures Versus Conventional Complete Dentures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Elgamal, Associate Professor of Prosthodontics, Mansoura University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R.25.11.82
Record Dates: First submitted 2025-12-03; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Swallowing Disorder
Keywords: complete denture; Fully digital; Food processing
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: This randomized crossover clinical trial evaluated swallowing function using the TOMASS test in patients fitted with 2 types of complete dentures (CDs): Conventionally fabricated CDS and Fully Digital fabricated CDs. Randomization process to participants was done to minimize the impact of the order of denture type on the measurements of swallowing threshold and Oral food processing assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventionally fabricated complete denture (Active Comparator): Each patient received two sets of dentures fabricated to identical functional and esthetic specifications, differing only in the manufacturing technique.
  The participants received conventional Complete dentures. Three months after denture use, the TOMASS test was done.
  Interventions: Procedure: Procedure for construction of complete denture either conventional or fully digital fabrication
- Fully digital fabricated complete denture (Active Comparator): Each patient received two sets of dentures fabricated to identical functional and esthetic specifications, differing only in the manufacturing technique.
  The participants received Fully digital fabricated complete denture. Three months after denture use, the TOMASS test was done.
  Interventions: Procedure: Procedure for construction of complete denture either conventional or fully digital fabrication

INTERVENTIONS:
Procedure: Procedure for construction of complete denture either conventional or fully digital fabrication — To ensure consistency and minimize patient visits, fabrication of both the conventional and fully digital complete dentures was conducted simultaneously during each clinical stage. All procedures were performed by the same prosthodontist, and efforts were made to standardize materials, occlusal schemes, and vertical dimension across both workflows for each patient.
  each patient received two sets of dentures fabricated to identical functional and esthetic specifications, differing only in the manufacturing technique.

SUMMARY:
The study aimed to compare the effects of fully digital versus conventional complete denture fabrication on oral food processing (mastication and swallowing of solids) in edentulous patients, using the Test of Mastication and Swallowing Solids (TOMASS).

In a randomized crossover study design was carried out on 14 completely edentulous participants (age 50-65 years, both sexes) in good general and oral health, each participants received two sets of dentures: one fabricated with conventional workflow (physical impressions, tooth arrangement, processing into heat polymerized acrylic) and one fully digital workflow (Intra-oral scanning , CAD/CAM design, 3D printed base and teeth,). Each denture was worn for 3 months; with a 2 week "wash out" period between wearing periods, during which participants reverted to their old dentures or no dentures. The order (Conventional complete denture first vs Digital complete denture first) was randomized. At the end of each denture period, Oral food processing performance was measured using TOMASS (solid cracker test): Swallowing threshold and TOMASS test parameters that include number of bites, number of masticatory cycles, number of swallows, and total time (from first bite to last swallow)

DETAILED DESCRIPTION:
Fourteen completely edentulous patients were participated in this study, their ages range from 50- 70 years. The participants were selected from Prosthodontics Department, Faculty of Dentistry, Mansoura University who are seeking for complete denture treatment. All participants will be completely edentulous for at least 6 months and have no previous experience with removable prosthesis. Subjects with temporomandibular joint disorders, head/neck injury, or with skeletal deformity were excluded from this study. All participants were Angel's class I maxillomandibular relation. Informed consent were written from each patient, and approval from the Faculty Ethical Committee will be obtained. The sample size was deter¬mined based on the number of chews for TOMASS test data from previous research. A computer software program (G*power, version 3.1.5, Kiel, Germany) was used for sample size calculation. 14 participants was detected with an effect size of 72%, 5% error probability, and 80% power.

Complete dentures construction:

At the first visit Direct intraoral scanning of both arches were performed with an intraoral scanner (TRIOS 3; 3Shape A/S). Cheek retractors were used to gently extend the movable soft tissues. The ridge crest were scanned first, followed by scans of the labial or buccal and palatal or lingual surfaces of the ridge. For the maxillary arch, the palate were additionally scanned. After establishing the overall contour in this manner, the remaining unscanned parts were scanned to finalize the complete arch scan. Subsequently, preliminary impressions were made with an irreversible hydrocolloid impression material.

At the second visit Definitive impressions will be made using auto-polymerizing acrylic resin custom tray. The tray will be traced using low fusing modeling green compound then zinc oxide eugenol impression will be taken. For the fabrication of conventional CDs, the record base will be fabricated with an auto-polymerizing acrylic resin. For the fabrication of digital CDs, the record base will be directly designed on the intraoral scan data by using a CAD software program (Dental System, v1.7.16.0; 3Shape A/S) and will be additively manufactured with a 3D-printing material (Next- Dent C&B; 3D Systems) and a 3D printer (NextDent 5100; 3D Systems). Following this, a wax occlusal rim were attached to the record base.

At the third visit Maxillo-mandibular relationship were recorded by using the record base and wax occlusal rim assembly with an occlusal relationship registration material for both groups, and appropriate artificial teeth will be selected. For the fabrication of digital CDs, the obtained inter-arch relationship were scanned with the intraoral scanner. Subsequently, the standard tessellation language (STL) files for both edentulous arches and the registered inter-arch relationship will be imported into a metrology software program (Geomagic Control X, v2018.0.1; 3D Systems). The maxillary portion in the STL file of the registered interarch relationship will be flipped normal, creating a new STL file, and the original maxillary edentulous STL file were superimposed over this new flipped file through a best-fit matching algorithm. The same procedure were followed with regard to the mandibular portion in the STL file of the registered inter-arch relationship. This procedure enabled accurate 3D orientation of the obtained intraoral scan data. Next, the border of the CDs will be set 1 mm shorter than the scan border within the CAD software program. The artificial teeth will be arranged virtually, and the trial dentures were additively manufactured with the3D-printing material (NextDent C&B; 3D Systems) and the 3D printer. For the conventional dentures the artificial teeth were arranged in the conventional manner.

At the fourth visit Trial dentures were evaluated in both groups. The procedure for preparing the definitive CDs were initiated after the participant had accepted the trial dentures. For the fabrication of digital CDs, the gingival portion and the artificial tooth portion were fabricated separately by using the 3D printer and 3D printing materials (NextDent Base and NextDent C&B; 3D Systems) and were subsequently attached to each other. Conventional CDs were fabricated by using flasking technique with long curing cycle.

At the fifth visit The predetermined CDs type were delivered and will be adjusted and follow up visits will be scheduled.

The participants were randomly allocated into two equal groups (7 per group). An independent examiner using a computer program, specifically Microsoft Excel, will carry out randomization process. The first group of 7 participants were received digital CDs. At 3 months after denture use, the TOMASS test were done. After 1 week washout period, the participants wearied the conventional CDs for an additional 3 months, then the TOMASS test will be repeated. The second group of 7 patients will initially receive conventional CDs. At three months after denture use, the TOMASS test will be done. Then after 1 week washout period the participants will receive the digital CDs, and the test will be repeated after an additional three months of denture use.

Oral processing assessment:

TOMASS test were utilized to assess participants' oral processing during ingestion of solid food. For this study, a commercially available cracker (biscuit) will be used. Participants will be instructed to sit on a chair in upright position and to eat the biscuit comfortably and as quickly as possible. They also will be asked to say their name out loud as it indicates that they had finished the test. Using a video recorder the procedure will be recorded for further analysis.

The recorded videos were then analyzed using the Avidemux 2.6 program to measure the following:

1. Swallowing threshold, which is the duration of chewing until the first swallow (determined by the moment of laryngeal elevation)
2. The TOMASS test parameters:

   1. Number of bites: The number of discrete bites taken to finish the cracker
   2. Number of masticatory cycles: As each cyclical mandibular movement up-down
   3. Number of swallows: As each vertical movement of the thyroid cartilage
   4. Total ingestion time: The time taken to complete the ingestion of the cracker from the first bite to the last.

ELIGIBILITY:
All participants were completely edentulous for at least 6 months,

* had no previous experience with removable prosthesis
* had Angel's class I maxillo-mandibular relation
* Willingness to comply with the study protocol and attending follow-up visits

Exclusion Criteria

* Participants with temporo-mandibular joint disorders.
* head/neck injury, or with skeletal deformity.
* Inability to wear dentures for extended periods or intolerance to the study

Ages: 50 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-11-17 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Swallowing threshold | 3 months after denture use
  Swallowing threshold, which is the duration of chewing until the first swallow (determined by the moment of laryngeal elevation)
The TOMASS test parameters: Number of bites: | 3 months after denture use
  Number of bites: The number of discrete bites taken to finish the cracker

SECONDARY OUTCOMES:
Number of masticatory cycles: | 3 months after denture use
  Number of masticatory cycles: As each cyclical mandibular movement up-down
Number of swallows | 3 months after denture use
  Number of swallows: As each vertical movement of the thyroid cartilage
Total ingestion time: | 3 months after denture use
  Total ingestion time: The time taken to complete the ingestion of the cracker from the first bite to the last.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Elgamal, Principal Investigator — Mansoura University; Abdallah M Ibrahim, Study Director — Mansoura University
Locations (1):
- Removable prosthodontics department,Faculty of dentistry,Mansoura university, #68 ElGomhoria Street, ElMansoura, Egypt. Mansoura, Eldakahlia, Egypt, 35516, Al Mansurah, Eldakahlia,, Egypt

IPD SHARING:
Plan to Share IPD: No